CLINICAL TRIAL: NCT03682198
Title: Neuro-Ox 2018: Assessment of Cerebral Oxygenation Under Three Clinically Relevant Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Sofie Pedersen, MD, Primary Investigator, University Hospital Bispebjerg and Frederiksberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Neuro-Ox 2018
Record Dates: First submitted 2018-08-28; First posted 2018-09-24 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Neurosurgery; Elective Craniotomy; General Anaesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One strategy for all enrolled patients: (Other): All patients will participate in three substudies, in which they also act as controls, with exposure to the same three interventions: 1) NIRS-measurement on skin, skull and dura, 2) Phenylephrine 0.1 mg iv., and 3) inspired oxygen fraction of 0.3 vs. 0.8
  Interventions: Device: NIRS measurements on skin, skull and dura; Drug: Phenylephrine's effect on brain oxygenation; Drug: Normal vs. high inspired oxygen

INTERVENTIONS:
Device: NIRS measurements on skin, skull and dura — During a neurosurgical procedure, we will measure the brain oxygenation with a NIRS-electrode, first on forehead skin, then on the skull and finally directly on dura.
Drug: Phenylephrine's effect on brain oxygenation — With a Clark-electrode (Licox(R)) in the white matter and a NIRS-electrode on the forehead skin, we will give a small dose (0.1 mg iv.) Phenylephrine.
Drug: Normal vs. high inspired oxygen — By the end of the neurosurgical procedure, still with a Clark-electrode in the white matter and a NIRS-electrode on forehead skin, we will change the inspired oxygen fraction from 0.3 to 0.8.

SUMMARY:
This is a prospective observational study, consisting of 3 substudies carried out during elective neurosurgery under general anaesthesia. Each participant will take part in all 3 substudies. First, the capability of Near Infra Red Spectroscopy (NIRS) to measure the brain oxygenation is examined. A NIRS-electrode is placed on forehead skin, on the skull, and on dura. Secondly, a small dose of Phenylephrine is given, and the brain oxygenation is measured by a Clark-electrode and a NIRS-electrode, to see how Phenylephrine affects these measurements. In the third substudy, the brain oxygenations' (NIRS and Licox) response to an inspired oxygen fraction of 0.30 vs. 0.80 is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) patients
* Elective craniotomy

Exclusion Criteria:

* Repeat craniotomy
* Preoperative hypotension (defined as systolic blood pressure below 110 mmHg)
* Preoperative hypoxia (defined as peripheral oxygen saturation (SpO2) < 90% without oxygen supplementation before surgery)
* No negative pregnancy test for women <50 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
ScO2 (NIRS-measured cerebral oxygen saturation) | During surgical procedure
  Difference in ScO2 between dura and skin (Primary analysis for substudy 1)

SECONDARY OUTCOMES:
PBrO2 (Partial pressure of brain tissue oxygen) | During surgical procedure
  Cerebral oxygenation, measured by a Clark-electrode (Licox (R)) (Primary outcome measure for substudy 2)
PBrO2 (Partial pressure of brain tissue oxygen) | 'Normoxia' is induced with FiO2 = 0.30 for 5 minutes, and then changed to 'Hyperoxia' with FiO2 = 0.80 for the subsequent 5 minutes, while registering the Licox-signal.
  Cerebral oxygenation during inspired oxygen fraction 0.80 vs. 0.30 (Primary outcome for substudy 3)
ScO2 (NIRS-measured cerebral oxygen saturation) | Measurements will be performed as the surgeon exposes the skull.
  Difference in ScO2 between dura and skull, and between skull and skin (this will be the secondary analyses of substudy 1)
ScO2 (NIRS-measured cerebral oxygenation) | NIRS signal is obtained continuously during the Phenylephrine intervention
  NIRS-signal during Phenylephrine intervention (this will be the secondary outcome of substudy 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark